CLINICAL TRIAL: NCT05844124
Title: A Comparison of Impacts of Different Exercise Programs on Individuals With Knee Pathology
Brief Title: Impact of Different Exercise Programs on Knee OA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Prakash Jayabalan MD, PhD, Director, Clinical Musculoskeletal Research, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00215669
Record Dates: First submitted 2023-02-06; First posted 2023-05-06 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis; Knee Osteoarthritis; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases
Keywords: Osteoarthritis; Knee; Knee Osteoarthritis Exercise
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases | interventions — Exercise; Control Groups

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The Principal Investigator will be masked to the patient treatment group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group: Standard of care land-based walking exercise (Active Comparator): Participants enrolled in the control group will be recommended national exercise recommendations pertianing to engaging in 150 minutes a week of moderate intensity exercise five times per week.
  Apart from these exercise sessions participants in this group will complete 3 separate evaluation sessions at the beginning, interim, and end of the study where they will be walking on a standard-of care treadmill for 30 minutes with blood draws at 0 and 30 minutes (only during beginning and end session), kinematic measure of gait parameters, measures of different cardiovascular parameters and cardiometabolic markers followed by thigh muscle strength testing.
  Interventions: Other: Exercise for Knee Osteoarthritis Recommendations (Control group)
- Intervention group 1: Lower-body positive-pressure supported low-load treadmill walking exercise (Experimental): Participants enrolled in the Lower-body positive-pressure (LBPP) supported low-load treadmill walking exercise will complete a total of two walking exercise sessions per week for a total of eight consecutive weeks (i.e. 16 exercise sessions in all). Each walking session will include 30-minute walking on a G-Trainer (AlterG Inc., Fremont, CA) under low-load walking conditions.
  Apart from these exercise sessions participants in this group will complete 3 separate evaluation sessions at the beginning, interim, and end of the study where they will be walking on a standard-of care treadmill for 30 minutes with blood draws at 0 and 30 minutes (only during beginning and end session), kinematic measure of gait parameters, measures of different cardiovascular parameters and cardiometabolic markers followed by thigh muscle strength testing.
  Interventions: Other: Exercise for Knee Osteoarthritis -(LBPP supported low-load treadmill Walking)
- Intervention group 2: Aquatic Walking exercise (Experimental): Participants enrolled in the aquatic exercise program will complete a total of two aquatic walking exercise sessions per week for a total of eight consecutive weeks (i.e. 16 exercise sessions in all). Each aquatic exercise program will include walking in the pool for 30 minutes at self-selected speeds under the guidance of an aquatic therapy instructor.
  Apart from these exercise sessions participants in this group will complete 3 separate evaluation sessions at the beginning, interim, and end of the study where they will be walking on a standard-of care treadmill for 30 minutes with blood draws at 0 and 30 minutes (only during beginning and end session), kinematic measure of gait parameters, measures of different cardiovascular parameters and cardiometabolic markers followed by thigh muscle strength testing.
  Interventions: Other: Exercise for Knee Osteoarthritis - (Aquatic Walking)

INTERVENTIONS:
Other: Exercise for Knee Osteoarthritis Recommendations (Control group) — Patients in this group will receive available exercise recommendations of 150 minutes of moderate intensity exercise per week (30 minutes per day).
  Arms: Control group: Standard of care land-based walking exercise
Other: Exercise for Knee Osteoarthritis -(LBPP supported low-load treadmill Walking) — Lower-body positive-pressure (LBPP) supported low-load treadmill walking exercise
  Arms: Intervention group 1: Lower-body positive-pressure supported low-load treadmill walking exercise
Other: Exercise for Knee Osteoarthritis - (Aquatic Walking) — Aquatic Walking exercise
  Arms: Intervention group 2: Aquatic Walking exercise

SUMMARY:
This study will examine and compare the changes in serum biomarkers, joint kinematics, and thigh muscle strength based on three different 8-week exercise protocols in individuals with knee pathology: Lower-body positive-pressure (LBPP) supported low-load treadmill walking and Aquatic exercise program and standard of care treadmill or community walking.

Investigators hypothesize that both the 8-week exercise programs which aim to partially off-load the knee joint will be associated with a significant reduction in serum biological markers of joint disease (tissue turnover, cartilage degradation and inflammation) in response to the exercise. The serum biological markers will be directly correlated to participant reported knee pain. Both the LBPP-supported low-load and the aquatic exercise regimens will result in significant increases in thigh muscle strength about the degenerative knee which in-turn will result in diminished knee pain and enhanced joint function. Investigators aim to compare these two exercise programs to understand if benefits of one far exceeds the other as compared to standard of care treadmill or community walking.

DETAILED DESCRIPTION:
The morphology and composition of healthy mature articular cartilage is optimized to its primary function of load transfer and distribution. In the osteoarthritic state however, homeostasis of the knee joint is significantly altered, such that as the load is placed on the joint there is a progressive worsening of cartilage damage over time. Altered joint mechanics and intra-articular biological processes are thought to play pivotal roles in the initial breakdown and potentiation of cartilage damage which is the hallmark finding in knee OA leading to knee pain. Aquatic therapy alleviates stress on joints and provides people with pain or arthritis a safe opportunity to engage in activity. Walking or running with weight support on a lower-body positive-pressure (LBPP) treadmill similar to aquatic exercise therapy is a novel training and rehabilitation modality for individuals with lower extremity pathologies due to its ability to limit pain. This treadmill provides a controlled off-loading of the lower extremities with significant benefit being shown after 12 weeks of training in overweight individuals with knee OA on knee pain, function and muscle strength. Although these methodologies (LBPP treadmill and aquatic therapy) alter the joint mechanics, the intra-articular biological effect on joint disease remains unknown.

Diminished muscle strength is a common symptom associated with onset of knee osteoarthritis. Quadriceps muscle impairment in patients with knee OA is well documented in the literature. Muscle impairments in patients with OA are not limited to quadriceps but also involve hamstrings. Muscle strength, especially quadriceps, is a major determinant of both performance-based and self-reported physical function in subjects with knee OA. The evidence supports the benefit of exercise therapy (both land and aquatic), including global and targeted resistance training, in reducing pain and improving function in subjects with knee OA however research to date has been unable to quantify the disease-modifying effect of any form of exercise.

A recent study from investigators laboratory in individuals with knee OA, walking at self-selected speed, found that at a single session of 45 minutes of 50% body weight (BW) walking on this treadmill leads to a significant decrease in knee joint pain, and reduced pathologic gait features. It also decreased the serum concentration of biomarkers of inflammation (IL-6 and IL-8), adipokines and cartilage tissue turnover (cartilage oligomeric matrix protein, COMP)24 compared to 100% full body weight walking. The benefits of both types of exercise are primarily as a result of the decreased effects of gravity with buoyancy or positive pressure being associated with decreased compressive and shear joint forces at the knee.25 To investigators' knowledge no prior study has performed a longitudinal clinical trial of either treatment in sedentary older individuals as a treatment for concurrent knee OA and CVD. The longitudinal use of such a treadmill may allow these individuals to safely engage in physical activity, reducing joint pain, improving function, and improving cardiovascular parameters. The present pilot study will establish the conditions and parameters for a future longer-term clinical trial that aims to compare of impacts of aquatic therapy exercise program and lower body positive pressure treadmill walking on biological markers of joint disease, joint kinematics and thigh muscle strength in individuals with knee pathology.

The study investigators propose is a randomized controlled trial in individuals with mild to moderate knee OA (n=15 in each group), evaluating the symptomatic, biochemical, and biomechanical benefits of 3 walking exercise treatments: 1) LBPP treadmill walking 2) aquatic walking 3) standard of care land-based or community walking exercise for the same duration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Diagnosis of unilateral or bilateral knee osteoarthritis
* Clinical AND/OR radiographic knee osteoarthritis.
* Clinical radiographic knee osteoarthritis: Symptoms of 2 or more knee pain, morning stiffness in the joint, crepitus on active movement, tenderness of the joint, bony enlargement of the joint, and lack of palpable warmth of the synovium
* Radiographic knee osteoarthritis: Kellgren-Lawrence score of 2 or greater using radiographs of the involved knee
* If the participant has had diagnostic radiographs within the previous 2 years at Shirley Ryan AbilityLab, we will use these previous radiographs to confirm diagnosis (these participants will complete a HIPAA authorization form so that we can access these images).
* If the participant has not had a diagnostic radiograph within the previous 2 years, the participant will complete a bilateral standing anteroposterior radiograph for the purpose of this study. These images are consistent with clinical care for diagnostic OA and minimally expose the individual to radiation (see attached form from radiology technician). All images taken as part of the study will be stored using the assigned study identifier, and therefore will not require any HIPAA authorization.
* Ability to walk without the use of aids (e.g., cane, walker)

Exclusion Criteria:

* Age < 50 years
* History of lower extremity total joint arthroplasty
* Current cardiovascular disease or hypertension that is uncontrolled
* History of neurological disorder that effects lower extremity function (i.e., stroke, peripheral neuropathy, multiple sclerosis, Parkinson's disease)
* Current ankle or hip pain
* Currently pregnant for female participants
* Weight over 400 lbs (181.4 kg), height less than 4'8" (142 cm) or over 6'4" (193 cm), 18.5" (47 cm) hip width, or 58" (147 cm) hip circumference

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain subscore on the Knee injury and Osteoarthritis Score (KOOS Survey) | Baseline, and 30 minutes of walking within session and also as a comparison between day 0, week 4, and week 8.
  Measured by the Pain Knee injury and Osteoarthritis Outcome Score subscale (KOOS subscales) as a comparison between different groups of the evolution of pain between Day 0 and Week 8. Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.

SECONDARY OUTCOMES:
Function | Baseline, and 30 minutes of walking within session and also as a comparison between day 0, week 4, and week 8
  Measured by the Function Knee injury and osteoarthritis score subscales (KOOS subscales) as a comparison between different groups of the evolution of function between Day 0 and Week 8.subscales) as a comparison between day 0, week 4, and week 8. Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
Symptoms | Baseline, and 30 minutes of walking within session and also as a comparison between day 0, week 4, and week 8
  Measured by the Symptoms Knee injury and Osteoarthritis Outcome Score subscales (KOOS subscales) as a comparison between different groups of the evolution of symptoms between Day 0 and Week 8.
Impact of Osteoarthritis on Quality of Life | Baseline, and 30 minutes of walking within session and also as a comparison between day 0, week 4, and week 8
  Measured by the Quality of life Knee injury and Osteoarthritis Outcome Score subscales (KOOS subscales). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
Change in Inflammatory cytokine (IL-6) concentration | Baseline, and 30 minutes of walking within session and also as a comparison between day 0 and week 8
  Serum (blood) marker concentration
Change in Inflammatory cytokine (IL-1B) concentration | Baseline, and 30 minutes of walking within session and also as a comparison between day 0 and week 8
  Serum (blood) marker concentration
Change in Inflammatory cytokine (IL-1RA) concentration | Baseline, and 30 minutes of walking within session and also as a comparison between day 0 and week 8
  Serum (blood) marker concentration
Questionnaire on Non-steroidal anti-inflammatory drugs (NSAID) use | Comparison between day 0, week 4, and week 8
  This questionnaire will include questions on participants' use of any pain medications and their frequency/dosage. The response will be recorded during pre, interim and post-evaluation sessions and will be studied for any changes.
Change in Inflammatory cytokine (IL-10) concentration | Baseline, and 30 minutes of walking within session and also as a comparison between day 0 and week 8
  Serum (blood) marker concentration
Six minute walk test | Comparison between day 0, week 4, and week 8
  Amount of distance walked in 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Jayabalan, MD, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No